CLINICAL TRIAL: NCT01896947
Title: Three Tesla Magnetic Resonance Imaging Compared to Magnetic Resonance Arthrogram in Diagnosing Superior Labrum Anterior Posterior (SLAP) Lesions
Brief Title: 3T MRI Versus MR Arthrogram in SLAP Lesions
Status: Withdrawn | Type: Observational
Why Stopped: Cost
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Stephanie Muh, MD, Staff Physician, Henry Ford Health System
Other Study IDs: SLAP MR study
Record Dates: First submitted 2013-07-08; First posted 2013-07-11 (Estimated); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Superior Labrum Anterior Posterior Lesion

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- MRI and MRA group: All patients will receive 3T MRI and MR arthrogram
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — evaluating to see if 3T MRI is as effective as MR arthrogram to diagnose labral pathology

SUMMARY:
The purpose of this study is to evaluate the diagnostic performance of three Tesla magnetic resonance imaging (3T MRI) compared to magnetic resonance arthrogram (MR arthrogram) in diagnosing superior labrum anterior posterior (SLAP) lesions. We hypothesize that 3T MRI will have non-inferior sensitivity compared to MR arthrogram in diagnosing SLAP lesions utilizing arthroscopy as our gold standard test. To evaluate our hypothesis, the investigators will include patients suspected to have a SLAP lesion on history and physical examination by a fellowship trained orthopaedic surgery. Patients will be offered advanced imaging (both 3T MRI and MR arthrogram) as well as arthroscopy for definitive diagnosis and treatment after consent is obtained. A fellowship trained musculoskeletal radiologist will perform and interpret the magnetic resonance tests while the arthroscopy will be performed by orthopaedic surgeons. The diagnostic characteristics of each imaging modality, including sensitivity, specificity, negative predictive value, and positive predictive value, will be compared to each other.

DETAILED DESCRIPTION:
Purpose: The purpose of this study is to evaluate the diagnostic performance of three Tesla magnetic resonance imaging (3T MRI) compared to magnetic resonance arthrogram (MR arthrogram) in superior labrum anterior posterior (SLAP) lesions.

Specific aims: 1) Determine the diagnostic performance of 3T MRI in SLAP lesions utilizing arthroscopy as the gold standard (2) Determine the diagnostic performance of MR arthrogram in SLAP lesions utilizing arthroscopy as the gold standard (3) Compare the diagnostic performance of 3T MRI and MR arthrogram in SLAP lesions in a non-inferiority trial

Rationale: SLAP lesions are difficult to diagnose, even with advanced imaging (1). MRI and MR arthrogram are imaging modalities used to diagnose SLAP lesions while arthroscopy is the gold standard for diagnosing SLAP lesions. Recent study indicates that 1.5T MRI is not suitable for diagnosing SLAP lesions due to low specificity (2). The sensitivity and specificity of MRI have been reported between 66-98% and 75-91%, respectively (3,4). The reported sensitivity and specificity of MR arthrogram is generally higher at 82-100% and 58-98%, respectively (5-8). However, because the MR arthrogram is an invasive diagnostic tool, both MR arthrogram and MRI are considered standards of practice in the evaluation of SLAP lesions. To the investigators' knowledge, no previous study of SLAP lesions has evaluated the performance of 3T MRI, which has better diagnostic capabilities compared to 1.5T MRI, and compared it to MR arthrogram.

Significance: By comparing the performance of the 3T MRI and MR arthrogram in diagnosing SLAP lesions, the investigators will be able to make important diagnostic recommendations. For example, if 3T MRI is non-inferior to MR arthrogram, then the discomfort, potential harm of contrast agents, and extra resources required for MR arthrogram could be avoided with a 3T MRI.

Subjects: Inclusion criteria are patients suspected to have a SLAP lesion, either in isolation or in combination with other shoulder pathology, on history and physical examination by a fellowship trained shoulder and elbow surgeon or fellowship trained sports surgeon. Furthermore, patients must be indicated for arthroscopy. As part of standard of care, included patients will provide consent for arthroscopic evaluation. Exclusion criteria include skeletally immature patients, previously diagnosed SLAP lesion, previous intervention for SLAP lesion, contrast dye allergy, and implants that are contra-indicated for MRI.

Project design and protocol: All patients meeting inclusion and exclusion criteria will be evaluated prospectively. Patients eligible for participation will be identified in the clinics of two fellowship trained orthopaedic surgeons. The surgeons will obtain consent for study participation as well as shoulder arthroscopy. Patients will subsequently be referred to the Department of Radiology for 3T MRI and MR arthrogram. Consent for a shoulder MR arthrogram will be obtained and performed by a fellowship trained musculoskeletal radiologist. MRI and MR arthrogram images will be read by a fellowship trained musculoskeletal radiologist. Each patient will then undergo shoulder arthroscopy and indicated interventions by fellowship trained orthopaedic surgeons.

Data Analysis: Specific Aim 1: Sensitivity, specificity, negative predictive value, and positive predictive values will be calculated for MRI utilizing arthroscopy as the gold standard. These calculations will be made from a 2x2 Table. Specific Aim 2: Sensitivity, specificity, negative predictive value, and positive predictive values will be calculated for MR arthrography utilizing arthroscopy as the gold standard. These calculations will be made from a 2x2 Table. Specific Aim 3: Sensitivity, specificity, negative predictive value, and positive predictive values will be compared for 3T MRI and MR arthrogram. The investigators will evaluate for non-inferiority of 3T MRI to MR arthrogram Descriptive statistics for the cohort will be calculated with mean, median, and frequencies and distributions reported as appropriate.

Justification for number of subjects: Based on the reported sensitivity and specificity of MRI and MR arthrogram in the literature, the study is estimated to be adequately powered at 30 patients for a non-inferiority trial.

Tentative schedule for completing the project: The investigators estimate that approximately ten patients per month will be eligible for this study, based on the practice patterns of the orthopaedic surgeons involved in this study. An additonal month will be required for data analysis and writing the report.

ELIGIBILITY:
Inclusion Criteria:

* SLAP lesion

Exclusion Criteria:

* Skeletally immature
* Previous SLAP lesion on ipsilateral side
* Implants contraindicated for MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All skeletally mature patients with a suspected SLAP lesion on clinical exam will be eligible for the study.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-09-29 (Actual); Primary Completion 2024-09-29 (Actual); Study Completion 2024-09-29 (Actual)

PRIMARY OUTCOMES:
Sensitivity 3T MRI | 3 months
Specificity 3T MRI | 3 months
Positive predictive value 3T MRI | 3 months
Negative predictive value 3T MRI | 3 months
Sensitivity MRA | 3 months
Specificity MRA | 3 months
Positive predictive value MRA | 3 months
Negative predictive value MRA | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Muh, MD, Principal Investigator — Henry Ford Hospital
Locations (1):
- Henry Ford Hospital, Detroit, Michigan, United States

REFERENCES:
- [Background] Chang D, Mohana-Borges A, Borso M, Chung CB. SLAP lesions: anatomy, clinical presentation, MR imaging diagnosis and characterization. Eur J Radiol. 2008 Oct;68(1):72-87. doi: 10.1016/j.ejrad.2008.02.026. Epub 2008 May 21. PMID 18499376
- [Background] Phillips JC, Cook C, Beaty S, Kissenberth MJ, Siffri P, Hawkins RJ. Validity of noncontrast magnetic resonance imaging in diagnosing superior labrum anterior-posterior tears. J Shoulder Elbow Surg. 2013 Jan;22(1):3-8. doi: 10.1016/j.jse.2012.03.013. Epub 2012 Aug 29. PMID 22938789
- [Background] Dinauer PA, Flemming DJ, Murphy KP, Doukas WC. Diagnosis of superior labral lesions: comparison of noncontrast MRI with indirect MR arthrography in unexercised shoulders. Skeletal Radiol. 2007 Mar;36(3):195-202. doi: 10.1007/s00256-006-0237-7. Epub 2006 Dec 1. PMID 17139503
- [Background] Connell DA, Potter HG, Wickiewicz TL, Altchek DW, Warren RF. Noncontrast magnetic resonance imaging of superior labral lesions. 102 cases confirmed at arthroscopic surgery. Am J Sports Med. 1999 Mar-Apr;27(2):208-13. doi: 10.1177/03635465990270021601. PMID 10102103
- [Background] Waldt S, Burkart A, Lange P, Imhoff AB, Rummeny EJ, Woertler K. Diagnostic performance of MR arthrography in the assessment of superior labral anteroposterior lesions of the shoulder. AJR Am J Roentgenol. 2004 May;182(5):1271-8. doi: 10.2214/ajr.182.5.1821271. PMID 15100131
- [Background] Applegate GR, Hewitt M, Snyder SJ, Watson E, Kwak S, Resnick D. Chronic labral tears: value of magnetic resonance arthrography in evaluating the glenoid labrum and labral-bicipital complex. Arthroscopy. 2004 Nov;20(9):959-63. doi: 10.1016/j.arthro.2004.08.017. PMID 15525929
- [Background] Bencardino JT, Beltran J, Rosenberg ZS, Rokito A, Schmahmann S, Mota J, Mellado JM, Zuckerman J, Cuomo F, Rose D. Superior labrum anterior-posterior lesions: diagnosis with MR arthrography of the shoulder. Radiology. 2000 Jan;214(1):267-71. doi: 10.1148/radiology.214.1.r00ja22267. PMID 10644135
- [Background] Jee WH, McCauley TR, Katz LD, Matheny JM, Ruwe PA, Daigneault JP. Superior labral anterior posterior (SLAP) lesions of the glenoid labrum: reliability and accuracy of MR arthrography for diagnosis. Radiology. 2001 Jan;218(1):127-32. doi: 10.1148/radiology.218.1.r01ja44127. PMID 11152790